CLINICAL TRIAL: NCT03427268
Title: A Phase II, Open-label, Multicentre Study of PM060184 in Patients With Advanced Colorectal Cancer After Standard Treatment.
Brief Title: Clinical Trial of PM60184 in Advanced Colorectal Cancer After Standard Treatment
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: PharmaMar (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PM60184-B-002-17
Record Dates: First submitted 2017-12-20; First posted 2018-02-09 (Actual); Results first posted 2021-05-24 (Actual); Last update posted 2021-05-24 (Actual); Status verified 2021-04

CONDITIONS: Advanced Colorectal Cancer
MeSH Terms: interventions — plocabulin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- PM060184 (Experimental): PM060184
  Interventions: Drug: PM060184

INTERVENTIONS:
Drug: PM060184 — PM060184: 9.3 mg/m2 PM060184 i.v. as a 30-minute infusion via a central or peripheral venous catheter.Dose can be rounded to the first decimal point.
  PM060184 will be administered on Day 1 and Day 8 q3wk. (Three weeks=one treatment cycle).

SUMMARY:
This trial will evaluate the efficacy of PM060184 in terms of progression-free survival at 12 weeks (PFS3) in advanced or metastatic Colorectal Cancer (CRC) patients with any KRAS mutation status (wild- type; mutated; or unknown status) progressing after standard treatments (fluoropyrimidine, irinotecan, and oxaliplatin).

Patients in this trial will receive PM060184 at a dose of 9.3 mg/m2 as a 30-minute intravenous (i.v.) infusion on Days 1 and 8 q3wk.

ELIGIBILITY:
INCLUSION CRITERIA:

1. Voluntarily written informed consent, obtained before the beginning of any study-specific procedures.
2. Age ≥ 18 years.
3. Histologically-cytologically documented adenocarcinoma of colon or rectum that has progressed to the last prior treatment before inclusion.
4. Measurable disease according to Response Evaluation Criteria in Solid Tumors (RECIST) v.1.1. If the only tumor lesion is situated in a previously irradiated area or in an area subjected to other loco-regional therapy, regression in the lesion must be demonstrated radiologically.
5. Previous treatment in any setting with fluoropyrimidine, oxaliplatin and irinotecan in any combination (unless any is contraindicated).

   1. Adjuvant chemotherapy-based treatments count as prior therapy, as long as relapse had occurred during or within six months of completion of such therapies.
   2. Cumulative dose of prior oxaliplatin (if any) must be known.
   3. Prior cetuximab, panitumumab, bevacizumab, aflibercept, and regorafenib are allowed.
6. No more than two prior therapies for metastatic disease.
7. Washout periods for prior therapies (defined in relation to planned start of study treatment [first dose administration]):

   1. At least three weeks since the last administration of an antineoplastic treatment (chemotherapy, biological, targeted or investigational therapies).
   2. At least three weeks since radiotherapy involving up to 35% of bone marrow (radiotherapy involving > 35% of bone marrow is not allowed) or two weeks since the end of palliative radiotherapy including single doses.
   3. At least four weeks since any major surgical procedure, open biopsy, or significant traumatic injury.
8. Eastern Cooperative Oncology Group (ECOG) performance status (PS) 0 or 1.
9. Life expectancy ≥ 3 months.
10. Adequate bone marrow, liver, and kidney function:

    1. Hemoglobin ≥ 9 g/dL.
    2. Absolute neutrophil count ≥ 1.5 × 109/L.
    3. Platelet count ≥ 100 × 109/L.
    4. Serum creatinine ≤ 1.5 mg/dL or calculated creatinine clearance ≥ 40 mL/min (Cockcroft-Gault formula).
    5. Albumin ≥ 2.5 g/dL.
    6. Total serum bilirubin ≤ 1.5 times the upper limit of normal (ULN), except in case of Gilbert syndrome.
    7. Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 3 × ULN (≤ 5.0 × ULN in the case of liver metastases).
11. Recovery to grade ≤ 1 from any toxicity due to previous therapy (including peripheral sensory/motor neuropathy but excluding alopecia).
12. Left ventricular ejection fraction (LVEF) by echocardiography (ECHO) or multiple-gated acquisition (MUGA) scan within normal range (according to institutional standards).
13. Evidence of non-childbearing status for women of childbearing potential (WOCBP). WOCBP must agree to use a highly effective contraceptive measure during the trial and up to six months after treatment discontinuation, and fertile male patients must agree to refrain from fathering a child or donating sperm during the trial and up to four months after treatment discontinuation.

EXCLUSION CRITERIA:

1. Prior exposure to PM060184.
2. Known hypersensitivity to the study drug class or study drug excipient in the formulation.
3. Patients with locally advanced disease amenable to local and/or curative therapy (surgery or radiotherapy) at study entry.
4. Other serious and/or relevant diseases or clinical situations that, in the opinion of the Investigator, are incompatible with the protocol (including any of the following):

   1. History of another neoplastic disease (except for basal cell carcinoma of the skin, superficial bladder tumors, or properly treated carcinoma in situ of the uterine cervix or melanoma in situ) unless in remission for at least five years and with no recurrence.
   2. Symptomatic cerebral and/or leptomeningeal metastasis, spinal cord compression or carcinomatous meningitis.
   3. Neuropathy of any etiology (other than that caused by previous antineoplastic therapy).
   4. History of cardiac disease, such as myocardial infarction, in the year prior to registration in the clinical trial; symptomatic/uncontrolled angina pectoris; congestive heart failure or uncontrolled cardiac ischemia; any type of uncontrolled arrhythmia, congenital and/or prolonged QT interval or abnormal LVEF, or uncontrolled arterial hypertension (according to the standards of the World Health Organization [WHO]).
   5. History of significant psychiatric disease.
   6. Active infection requiring antibiotic, antifungal or antiviral treatment that, in the opinion of the Investigator, could compromise the patient's capacity to tolerate the therapy.
   7. Known active liver (hepatitis B or C or cirrhosis) or renal disease.
   8. Known human immunodeficiency virus (HIV) infection.
   9. Any other concomitant pathology that could jeopardize the patient's safety or commitment to complete the clinical trial.
   10. Inability or refusal to comply with the protocol or with the clinical trial procedures.
5. Pregnancy or lactation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2018-01-16 (Actual); Primary Completion 2019-02-11 (Actual); Study Completion 2019-02-11 (Actual)

CONTACTS AND LOCATIONS:
Locations (5):
- US017, Los Angeles, California, United States
- CA001, Toronto, Ontario, Canada
- Spain (3):
  - ES001, Barcelona
  - ES009, Madrid
  - ES002, Valencia

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The first informed consent was signed on 16 January 2018 and the first study treatment administration was on 8 February 2018. The cutoff date for the results was 11 February 2019 (date of last follow-up).
Groups:
- PM060184: PM060184 was administered i.v. via a central line or a peripheral venous catheter (in 30-min administration) at a dose of 9.3 mg/m2 on Day 1 and Day 8 every three weeks (q3wk) (three weeks = one treatment cycle) (dose can be rounded to the first decimal point).
Period: Overall Study
Arm/Group | PM060184
Started | 32
Completed | 0
Not Completed | 32
Not completed — Progressive disease | 25
Not completed — Never treated | 2
Not completed — Compassionate use | 1
Not completed — Withdrawal by Subject | 1
Not completed — Adverse Event | 3

BASELINE CHARACTERISTICS:
Arm/Group | PM060184
Number analyzed (Participants) | 32
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 23
  >=65 years | 9
Age, Continuous [Median (Full Range); unit: years] | 62 [36 to 74]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17
  Male | 15
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 32
Region of Enrollment [Count of Participants; unit: Participants]
  Canada | 1
  Spain | 31
Eastern Cooperative Oncology Group Performance Status [Count of Participants; unit: Participants] — PS 0 Fully active able to carry on all pre-disease performance without restriction PS 1 Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature PS 2 Ambulatory and capable of all selfcare but unable to carry out any work activities up and about more than 50% of waking hours PS 3 Capable of only limited selfcare confined to bed or chair more than 50% of waking hours PS 4 Completely disabled cannot carry on any selfcare; totally confined to bed or chair PS 5 Dead
  Participants
    PS 0 | 15
    PS 1 | 17
Stage at diagnosis [Count of Participants; unit: Participants] — 0:Only in mucosa/inner lining I:Into mucosa/muscular layer. Not into nearby tissue (NT)/lymph nodes (LN) IIA:Into wall. Not into NT/LN IIB:Into layers of muscle to lining of abdomen. Not to nearby LN IIC:Into wall and into nearby structures. Not to nearby LN IIIA:Into inner lining/muscle layers of intestine. Not into other body parts IIIB:Into bowel wall or to surrounding organs and into 1-3 LN or to a nodule of tumor in tissues but not in LN. Not in other body parts IIIC:4+ LN. Not to other body parts IVA:1 distant part of body IVB:>1 part of body IVC:Into peritoneum
  Participants
    Stage I | 1
    Stage IIIB | 5
    Stage IIIC | 2
    Stage IV | 17
    Stage IVA | 3
    Stage IVB | 3
    UK | 1
Primary tumor side [Count of Participants; unit: Participants]
  Left | 22
  Right | 10
Histology grade at diagnosis [Count of Participants; unit: Participants]
  G1: Well differentiated | 8
  G2: Moderately differentiated | 18
  G4: Undifferentiated | 1
  GX: Grade cannot be assessed | 5
KRAS mutation status [Count of Participants; unit: Participants]
  Mutated | 25
  Not done | 6
  Unknown | 1
Sites involved [Count of Participants; unit: Participants]
  1 site | 5
  2 sites | 12
  3 sites | 8
  4 sites | 5
  6 sites | 1
  7 sites | 1
Peripheral neuropathy [Count of Participants; unit: Participants]
  Yes | 19
  No | 13
Prior surgery [Count of Participants; unit: Participants]
  Yes | 28
  No | 4
Prior radiotherapy [Count of Participants; unit: Participants]
  Concurrent | 1
  Palliative | 4
  No | 27
Prior anticancer lines [Count of Participants; unit: Participants]
  1 line | 1
  2 lines | 26
  3 lines | 5
Best response to last prior therapy [Count of Participants; unit: Participants] — CR, complete response: disappearance of all lesions; PD, disease progression: ≥10% increase in target lesion size and does not meet tumor density criteria of PR density; PR, partial response: ≥10% decrease in target lesion size or ≥15% decrease in tumor density; SD, stable disease: none of the CR, PR, or PD criteria met; UK,unknown
  Participants
    CR | 2
    PR | 3
    SD | 14
    PD | 9
    UK | 4
Weight [Median (Full Range); unit: Kg] | 67 [39.6 to 105.5]
Height [Median (Full Range); unit: cm] | 166 [150 to 183]
Body surface area [Median (Full Range); unit: m^2] | 1.8 [1.3 to 2.3]
Time from diagnosis of advanced disease to study entry [Median (Full Range); unit: months] | 17.3 [5.8 to 69.5]
Time from first diagnosis to first PM060184 infusion [Median (Full Range); unit: months] | 22.9 [7.9 to 57.1]
Time from prior last progression before study entry [Median (Full Range); unit: months] | 1.2 [0 to 3.2]
Time from stop date of prior chemotherapy to study entry [Median (Full Range); unit: months] | 1.8 [0.1 to 6.3]

OUTCOME MEASURES:

1. Primary Outcome: Progression-free Survival Rate at Three Months
Description: Progression-free survival rate at 12 weeks (PFS3), defined as the rate estimate of the percentage of patients who are alive and progression-free at 12 weeks (~3 months) after the first treatment administration. Progression is defined using Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0), as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions
Time Frame: Time from the first day of study treatment to the day of assessment of progression, death or last tumor evaluation, up to 3 months
Population: 2 patients were never treated; 1 treated patient not receive 2 administrations over 2 cycles.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | PM060184
Number analyzed (Participants) | 29
percentage of participants | 20.7 [8 to 39.7]

2. Secondary Outcome: Overall Survival (OS)
Description: Overall Survival (OS), defined as the time from the first day of treatment to the date of death or last contact.
Time Frame: From the first day of treatment to the date of death or last contact, up to 12 months
Population: 2 patients were never treated; 1 treated patient not receive 2 administrations over 2 cycles
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | PM060184
Number analyzed (Participants) | 29
months | 9.8 [4.6 to NA] — not reached

3. Secondary Outcome: Progression Free Survival (PFS)
Description: Progression-free survival (PFS), defined as the time from the first day of study treatment to the day of assessment of progression, death or last tumor evaluation. Progression is defined using Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0), as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions.
Time Frame: Time from the first day of study treatment to the day of assessment of progression, death or last tumor evaluation, up to 12 months
Population: 2 patients were never treated; 1 treated patient not receive 2 administrations over 2 cycles
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | PM060184
Number analyzed (Participants) | 29
months | 2.6 [1.3 to 2.8]

4. Secondary Outcome: Overall Response Rate (ORR)
Description: Overall Response Rate defined as the percentage of patients with either complete response (CR) or partial response (PR) according to RECIST v.1.1.
  CR, complete response: disappearance of all lesions; PD, disease progression: ≥10% increase in target lesion size and does not meet tumor density criteria of PR density; PR, partial response: ≥10% decrease in target lesion size or ≥15% decrease in tumor density; SD, stable disease: none of the CR, PR, or PD criteria met; RECIST, Response Evaluation Criteria in Solid Tumors
Time Frame: as for outcome 3
Population: 2 patients were never treated; 1 treated patient not receive 2 administrations over 2 cycles
Measure: Count of Participants; unit: Participants
Arm/Group | PM060184
Number analyzed (Participants) | 29
Participants
  SD <3 months | 9
  SD ≥3 months | 7
  PD | 13

ADVERSE EVENTS:
Time Frame: Patients were assessed between study start date and study completion date, approximately 1 year
Description: Patient excluded for analysis of safety: Two patients were never treated
Arm/Group | PM060184
All-Cause Mortality (participants affected / at risk) | 16/30
Serious Adverse Events (participants affected / at risk) | 6/30
Other Adverse Events (participants affected / at risk) | 30/30
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PM060184 (N=30)
Alanine aminotransferase increased (Investigations) | 3 (3)
Aspartate aminotransferase increased (Investigations) | 3 (3)
Blood bilirubin increased (Investigations) | 1 (1)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1)
Pyrexia (General disorders) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 1 (1)
Pneumonia pneumococcal (Infections and infestations) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PM060184 (N=30)
Deep vein thrombosis (Vascular disorders) | 2 (7)
Hypertension (Vascular disorders) | 2 (9)
Alanine aminotransferase increased (Investigations) | 2 (2)
Aspartate aminotransferase increased (Investigations) | 3 (3)
Blood bilirubin increased (Investigations) | 3 (5)
Gamma-glutamyltransferase increased (Investigations) | 2 (2)
Platelet count decreased (Investigations) | 2 (2)
Weight decreased (Investigations) | 3 (7)
Anaemia (Blood and lymphatic system disorders) | 7 (14)
Neutropenia (Blood and lymphatic system disorders) | 3 (3)
Dysaesthesia (Nervous system disorders) | 3 (10)
Dysgeusia (Nervous system disorders) | 2 (4)
Hypoaesthesia (Nervous system disorders) | 3 (9)
Neurotoxicity (Nervous system disorders) | 2 (7)
Paraesthesia (Nervous system disorders) | 14 (52)
Peripheral sensory neuropathy (Nervous system disorders) | 3 (12)
Asthenia (General disorders) | 22 (74)
Chest pain (General disorders) | 2 (4)
Pyrexia (General disorders) | 5 (10)
Anxiety (Psychiatric disorders) | 2 (7)
Insomnia (Psychiatric disorders) | 2 (9)
Abdominal distension (Gastrointestinal disorders) | 2 (2)
Abdominal pain (Gastrointestinal disorders) | 20 (66)
Abdominal pain upper (Gastrointestinal disorders) | 5 (15)
Constipation (Gastrointestinal disorders) | 19 (61)
Diarrhoea (Gastrointestinal disorders) | 11 (33)
Nausea (Gastrointestinal disorders) | 9 (23)
Vomiting (Gastrointestinal disorders) | 4 (7)
Alopecia (Skin and subcutaneous tissue disorders) | 14 (54)
Pruritus (Skin and subcutaneous tissue disorders) | 2 (11)
Arthralgia (Musculoskeletal and connective tissue disorders) | 5 (13)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 2 (6)
Decreased appetite (Metabolism and nutrition disorders) | 10 (26)
Device related infection (Infections and infestations) | 2 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The only disclosure restriction on the PI is that the sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period that is more than 60 days but less than or equal to 180 days from the time submitted to the sponsor for review.

DOCUMENTS (2):
  • Study Protocol (2017-07-27): https://cdn.clinicaltrials.gov/large-docs/68/NCT03427268/Prot_000.pdf
  • Statistical Analysis Plan (2018-02-20): https://cdn.clinicaltrials.gov/large-docs/68/NCT03427268/SAP_001.pdf